CLINICAL TRIAL: NCT03177447
Title: ENABLE: CHF-PC (Educate, Nurture, Advise, Before Life Ends: Comprehensive Heartcare for Patients and Caregivers)
Brief Title: ENABLE: CHF-PC (Comprehensive Heartcare For Patients and Caregivers)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Palliative Care Research Center (Other)
Responsible Party: Principal Investigator, Marie Anne Bakitas, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: X130827010
Record Dates: First submitted 2017-05-09; First posted 2017-06-06 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure, Congestive
Keywords: Cardiac Failure; Congestive Heart Failure; Heart Decompensation; Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Summative evaluation trial of ENABLE CHF-PC (Other): Single arm summative evaluation study was selected for several reasons: 1) to continue to determine recruitment feasibility; 2) retention- our prior work has demonstrated fairly equal dropouts in the intervention and control conditions, hence we believe we will be able to judge retention in a single arm design; 3) using a small randomized controlled trial (RCT) for power estimates runs a high risk of either overestimating or underestimating treatment effects; and 4) most importantly, the primary purpose of this study is to determine intervention efficacy. Therefore delivering the intervention to the maximum number of participants given the limitations of 2-year pilot funding allows the investigators to obtain the maximal input and experience with the intervention that is needed to achieve the study's Aim 1.
  Interventions: Behavioral: ENABLE CHF-PC

INTERVENTIONS:
Behavioral: ENABLE CHF-PC — An Advanced Practice Palliative Care Nurse Coach implements Charting Your Course (CYC), a phone-based, 6-session patient curriculum and a 3-session caregiver curriculum, followed by monthly phone supportive care follow-up. Sessions 1-3 incorporate Hegel's problem-solving approach that was modified to counsel seriously ill patients using MacMillan's COPE model reactivity, which includes 4 components: Creativity, Optimism, Planning and Expert information. These sessions address adjusting to chronic illness, symptom management, communication, and decision-making. Patient sessions 4-6 comprise OUTLOOK, a life review intervention to improve QOL in serious illness developed at Duke.

SUMMARY:
Background: Early palliative care (EPC) is recommended but rarely integrated with advanced heart failure (HF) care. This pilot study engaged patients and family caregivers to study the feasibility and site differences in a two-site EPC trial, ENABLE CHF-PC (Educate, Nurture, Advise, Before Life Ends Comprehensive Heartcare for Patients and Caregivers).

An EPC feasibility study (4/1/14-8/31/15) was conducted for patients with New York Heart Association (NYHA) Functional Class III/IV HF and their caregivers in academic medical centers in the northeast and southeast U.S. The EPC intervention comprised: 1) an in-person palliative care consultation; and 2) telephonic nurse coach sessions and monthly calls. Patient- and caregiver-reported outcomes were collected for quality of life (QOL), symptom, health, anxiety, and depression outcomes at baseline, 12- and 24-weeks. Linear mixed-models were used to assess baseline to week 24 longitudinal changes. The intervention was tailored to rural, older adults (age≥65) with advanced HF in reducing HF morbidity and improving patient and caregiver QOL and quality of care.

DETAILED DESCRIPTION:
High quality trials have demonstrated positive patient and family caregiver outcomes from early palliative care (EPC) in cancer However, given the difficulties in prognostication, the prevalence of sudden cardiac death, and an erratic illness trajectory, it is not clear when or how to integrate palliative care in HF. Furthermore, the high morbidity and mortality of HF in persons with low income, poor education, minority race, and residence in rural, medically-underserviced areas further complicates appropriate timing of integration.

To address these challenges, patients and family members were actively engaged to aid in the development of ENABLE CHF-PC (Educate, Nurture, Advise, Before Life Ends Comprehensive Heartcare for Patients and Caregivers), a telephonic EPC intervention for rural-dwelling, underserved HF patients and their family caregivers. In a proof-of-concept, formative evaluation study, materials and protocols were translated from our successful EPC ENABLE oncology model to a HF population. This study demonstrated acceptability, feasibility, and a signal of potential efficacy in an educationally, socioeconomically, and racially homogeneous sample of 11 patient-caregiver dyads. Thus, the current ENABLE CHF-PC feasibility trial was conducted in a northeastern and a southeastern US academic center to capture the perspectives of a more demographically and culturally-diverse sample. The purpose of this study was to: 1) determine the feasibility of recruiting and retaining patient-caregiver dyads for 24 weeks in a rural, racially-diverse sample and 2) explore longitudinal patient and caregiver outcomes including QOL, global health, anxiety, and depression to inform intervention and protocol modifications for a larger clinical efficacy trial.

Study Design: In this feasibility study, conducted April 1, 2014 to December 31, 2015, individuals with American College of Cardiology (ACC) /American Heart Association (AHA) Class C/D and/or NYHA Stage III/IV HF and their family caregivers received the ENABLE CHF-PC intervention and were followed for 24 weeks. The study protocol was approved by the institutional review boards of Dartmouth College (Lebanon, New Hampshire) and the University of Alabama at Birmingham (Birmingham, Alabama).

Setting and Sample: Study participants were recruited from cardiology clinics at Dartmouth-Hitchcock Medical Center (DHMC) and the University of Alabama at Birmingham (UAB). Study coordinators at both sites reviewed outpatient cardiology clinic schedules to identify eligible patients. Following physician approval, a study coordinator approached patients and their caregivers during a clinic appointment to explain the study and obtain consent.

Data Collection and Measures: Study coordinators completed measures with patients and caregivers by phone at baseline, 12- and 24-weeks. Baseline demographics included age, gender, race/ethnicity, religion, marital and work status, educational level, and medical insurance. Clinical characteristics abstracted from electronic health records included NYHA class, ejection fraction, presence of an implanted heart device, medications, and laboratory data. These data were entered into the Seattle Heart Failure Model (SHFM) a web-based calculator to compute 1-, 2- and 5-year survival estimates https://depts.washington.edu/shfm/). Nurse coaches also informed patients and caregivers that the purpose of this pilot trial was to determine acceptability in a new population - patients with heart failure from 2 distinctly different regions/cultures. Nurses recorded sessions, and tracked patient and caregiver feedback on intervention components that were found to be helpful or in need of improvement.

Statistical Analysis: The feasibility primary aim was determined by monitoring study status (enrolled, deceased, lost to follow-up) and calculating intervention and measurement completion (e.g. actual # completed/possible # per protocol). Patient and caregiver demographic characteristics were tabulated and compared between sites with bivariate tests of association and effect sizes (Cohen's d or d-equivalent or nominal variables). Associations were assessed between baseline characteristics and participant attrition using simple logistic regressions. Estimated odds ratios were used to determine associations between patient characteristics and attrition.

Longitudinal, fitted, linear mixed methods, adjusted for covariates associated with attrition were used to estimate participant-reported outcomes' changes from baseline to follow-up (12-week and 24-week means combined). Change estimates were transformed to effect sizes (Cohen's d) using baseline estimates of pooled standard deviations. Change was estimated overall and by site. All analyses were conducted using SAS v9.4.

Due to the exploratory nature of the study, the analysis relied on effect size estimation using Cohen's guidelines for magnitude of effect size d (i.e. small: 0.2, moderate: 0.5, and large: 0.8) rather than hypothesis testing to interpret results; however p-values are also provided for completeness.

ELIGIBILITY:
Patient Inclusion Criteria:

1. English-speaking and able to complete baseline interview
2. Age ≥65 (Age criteria was reduced to ≥50 y/o given regional experience with HF population)
3. NYHA Stage III/IV heart failure; American College of Cardiology (ACC) Class C/D
4. Have a land-based phone or reliable cellular phone service
5. Have an agreeable partner willing to participate in the study* (recommended) *In our previous studies we have not required patients to have a care partner for eligibility. In this study it is essential that we have an adequate number of caregivers to test the caregiver intervention. Therefore patients without a care partner will still be considered but the final study sample size may need to be adjusted to ensure an adequate caregiver sample.

Patient Exclusion Criteria:

1. Non-correctable hearing loss
2. Dementia or significant confusion (as measured by a Callahan score of ≤3
3. Diagnostic and Statistical Manual (DSM) -IV Axis I diagnosis (e.g. schizophrenia, bipolar disorder) or active substance use disorder

Caregiver Inclusion Criteria:

1. "Caregiver" is identified by the patient as "a person who knows you well and is involved in your medical care". May be a spouse or adult family member or friend living in the same household or considered by the patient to be the primary caregiver and be willing to participate."
2. English-speaking and able to complete baseline interview 3. Have a land-based phone or reliable cellular phone service.

Caregiver Exclusion Criteria:

1. Non-correctable hearing loss.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment for a large-scale RCT. | From Date of Enrollment to 24 Weeks
  Number (#) of participants enrolled within 2 years compared to study's target goal.
Feasibility of retention for a large-scale RCT. | From Date of Enrollment to 24 Weeks
  Number (#) of participants completing study activities by 24 weeks.
Feasibility of intervention completion for a large-scale RCT. | From Date of Enrollment to 24 Weeks
  Number (#) of participants completing all intervention sessions by 24 weeks.
Feasibility of measurement completion for a large-scale RCT. | From Date of Enrollment to 24 Weeks
  Number (#) of participants completing outcomes measures by 24 weeks.

SECONDARY OUTCOMES:
Patient Quality of Life | Baseline, week 12, and week 24.
  Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered HF-specific questionnaire that describes physical limitations (1 item), symptoms (frequency-4 items,severity-3 items, change over time-1 item) self-efficacy/ knowledge (2 items), social interference (1 item) and QOL (3 items). Individual domains show high internal consistency reliability (Cronbach's alpha's .62-.90). It is reported to take 6 minutes to complete. Two summary scores (functional and clinical) can be calculated. It is reported to be more sensitive to clinical change than other HF-specific measures. Scores range from 0-100 wherein higher scores indicate better health status.
Patient Quality of Care | Baseline, week 12, and week 24.
  Patient Assessment of Chronic Illness Care (PACIC) is a 20-item patient reported measure of chronic illness care (CIC) health counseling behaviors. It consists of the five CIC constructs: patient activation, delivery system/ decision support, goal setting, problem-solving, and follow-up/ coordination. It has good internal consistency with Cronbach alphas ranging from .78 to .90, and test-retest reliability, estimated by intracluster correlation coefficient (ICC), was at least 0.77.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Bakitas, DNSc, NP-C, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dartmouth-Hitchcock Medical Center, Dartmouth College, Dartmouth-Hitchcock Heart & Vascular Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Bakitas M, Dionne-Odom JN, Pamboukian SV, Tallaj J, Kvale E, Swetz KM, Frost J, Wells R, Azuero A, Keebler K, Akyar I, Ejem D, Steinhauser K, Smith T, Durant R, Kono AT. Engaging patients and families to create a feasible clinical trial integrating palliative and heart failure care: results of the ENABLE CHF-PC pilot clinical trial. BMC Palliat Care. 2017 Aug 31;16(1):45. doi: 10.1186/s12904-017-0226-8. PMID 28859648